CLINICAL TRIAL: NCT04362163
Title: Study for Testing and Reviewing Improvised PPE Effectiveness 3 (STRIPE-3) - a Third Comparative Trial Assessing the Safety of Improvised PPE
Brief Title: Study for Testing and Reviewing Improvised PPE Effectiveness 3 (STRIPE-3)
Acronym: STRIPE-3
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: TAP_PRG_21_04_2020_2
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: Personal protective equipment

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Snorkel-based improvised personal protective equipment — An improvised PPE design based on a full face snorkel mask mated to a heat-and-moisture exchange filter via a 3D printed adaptor.

SUMMARY:
Personal protective equipment (PPE) is vital to ensuring staff safety during the COVID-19 pandemic. Properly designed, formal PPE (fPPE) is in increasingly short supply, and a series of improvised PPE (iPPE) designs have been widely circulated on the internet, particularly on social media. Groups have started to publicise these devices through websites and the lay press. Some are even using crowd-funding to finance the purchase of these systems with the intention of supplying NHS workers in place of approved systems.

It is not clear what degree of testing these systems have undergone. The investigators are already planning trials formally investigating the quality of seal offered by these improvised systems. Currently the team are investigating a designed based on a modified snorkel mask (STRIPE-1). In the current study the investigators wish to extend this investigation to consider the atmosphere within the mask.

This is an important question, as modifications to the snorkel design have changed the way gases mix within the system. This might increase the risk that the user will rebreathe expired gases, which will dilute the amount of oxygen available to them, and increase the carbon dioxide levels to which they are exposed. At extreme deviations, these might pose a potential health hazard over and above the risks posed by COVID-19 exposure via a poor mask seal.

This study will therefore recruit a convenience sample of 10, and request they wear two masks sequentially. These masks will comprise: a formally designed and tested commercial FFP3 mask, and one design of improvised PPE, based on the snorkel design available on the internet.

Each mask will be worn for a total of 40 minutes. In the first 20 minutes measurements will be taken with the user at rest. In the second 20 minutes measurements will be taken while the user undertakes light exercise.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Healthy adults, male or female, aged 18 or more
* Clean-shaven at the point of testing
* Willing and able to undertake 20 minutes of light exercise e.g. stepping

Exclusion Criteria:

* They have facial hair that would disrupt the seals of the mask
* They have significant facial injuries or malformations that preclude a good mask seal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruits will be drawn from amongst staff at Guy's and St Thomas' NHS Foundation Trust (London, UK) who are required to be fit-tested on tight-fitting FFP3 masks as part of their normal clinical duties.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Oxygen concentration while wearing purpose-designed mask | 40 minutes starting from intervention (donning of mask)
  5-minute measurement of oxygen concentration in inspired and expired gases
Oxygen concentration while wearing improvised snorkel-based mask | 40 minutes starting from intervention (donning of mask)
  5-minute measurement of oxygen concentration in inspired and expired gases

SECONDARY OUTCOMES:
Carbon dioxide concentration while wearing purpose-designed mask | 40 minutes starting from intervention (donning of mask)
  5 minute measurement of carbon dioxide concentration in inspired and expired gases
Carbon dioxide concentration while wearing improvised snorkel-based mask | 40 minutes starting from intervention (donning of mask)
  5 minute measurement of carbon dioxide concentration in inspired and expired gases
Heart rate while wearing purpose-designed mask | 40 minutes starting from intervention (donning of mask)
  5 minute measurement of heart rate
Heart rate while wearing improvised snorkel-based mask | 40 minutes starting from intervention (donning of mask)
  5 minute measurement of heart rate
Respiratory rate while wearing purpose-designed mask | 40 minutes starting from intervention (donning of mask)
  5 minute measurement of respiratory rate
Respiratory rate while wearing improvised snorkel-based mask | 40 minutes starting from intervention (donning of mask)
  5 minute measurement of respiratory rate
Oxygen saturation while wearing purpose-designed mask | 40 minutes starting from intervention (donning of mask)
  5 minute measurement of oxygen saturation
Oxygen saturation while wearing improvised snorkel-based mask | 40 minutes starting from intervention (donning of mask)
  5 minute measurement of oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Greig, MBChB, Study Chair — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No